CLINICAL TRIAL: NCT00006212
Title: Phase I Study of Interstitial Colloidal 32P Integrated With External Radiation Therapy and Chemotherapy in the Treatment of Non-Resectable or Medically Inoperable Non-Small Cell Carcinoma of the Lung
Brief Title: Phosphorus-32 Plus Radiation Therapy and Chemotherapy in Treating Patients With Stage II or Stage III Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Center for Molecular Medicine (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067812; CMM-99003; NCI-V00-1586
Record Dates: First submitted 2000-09-11; First posted 2004-05-26 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-02

CONDITIONS: Lung Cancer
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Vinblastine; Phosphorus-32; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: vinblastine sulfate
Radiation: phosphorus P32
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as phosphorus-32 may make the tumor cells more sensitive to radiation therapy. Chemotherapy combined with radiation therapy and phosphorus-32 may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of phosphorus-32 plus radiation therapy and chemotherapy in treating patients who have stage II or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dosimetry and toxicity of interstitial phosphorus P32 colloid plus chemotherapy and radiotherapy in patients with previously untreated stage II, IIIA, or IIIB non-small cell lung cancer. II. Determine the maximum tolerated dose of phosphorus P32 colloid in these patients. III. Determine the response in patients treated with this regimen.

OUTLINE: This is a dose escalation study of phosphorus P32 colloid. Patients receive vinblastine IV on days 1, 8, 15, 22, and 29; cisplatin IV over 30-60 minutes on days 1 and 29; and phosphorus P32 colloid interstitially on day 50. Patients with tumor size less than 8.0 cm receive radiotherapy following phosphorus P32 injection 5 days a week for 6.5 weeks. Patients with tumor size greater than 8.0 cm receive radiotherapy 5 days a week for 4.5 weeks prior to phosphorus P32 injection, and for an additional 2.5 weeks following injection. Cohorts of 3 patients receive escalating doses of phosphorus P32 colloid until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicity. Patients are followed every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed, previously untreated stage II, IIIA, or IIIB non-small cell lung cancer Unresectable or inoperable disease OR Refusal of surgery Tumor reachable by CT guided needle placement Bidimensionally measurable disease by chest x-ray or CT scan No clinical/radiographic evidence of metastatic disease

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Neutrophil count at least 1,900/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (transfusion allowed) Hepatic: Adequate hepatic function Renal: BUN no greater than 25 mg/dL Creatinine no greater than 1.5 mg/dL Other: Less than 5% weight loss Able to receive induction chemotherapy No second malignancy within the past 5 years except skin cancer Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to thorax Surgery: See Disease Characteristics No prior resection at primary site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11

CONTACTS AND LOCATIONS:
Overall Officials: Wayne S. Court, MD, PhD, Study Chair — Center for Molecular Medicine
Locations (1):
- Center for Molecular Medicine, Garden City, New York, United States